CLINICAL TRIAL: NCT05699902
Title: The Effect of Pectoral Nerve Block as a Part of Enhanced Recovery After Mastectomy
Brief Title: Pectoral Nerve Block During Mastectomy
Acronym: PNB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Salah Abd-Ellah, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pectoral nerve block in breast
Record Dates: First submitted 2022-12-11; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer Female; Pain, Postoperative
Keywords: Breast cancer; Pain after mastectomy; PECs block
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Interventional
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECs block group (Active Comparator): Female undergone mastectomy and received pectoral nerve block
  Interventions: Procedure: PECs block during mastectomy
- Non PECs block group (Sham Comparator): Female undergone mastectomy and not received pectoral nerve block but have received conventional analgesic methods
  Interventions: Procedure: Sham block

INTERVENTIONS:
Procedure: PECs block during mastectomy — The patients were randomised to receive a PECS block consisting of 30 ml of levobupivacaine 0.25% after induction of anaesthesia (PECS group) or a saline mock block (control group). The patients answered a 40-item QoR questionnaire (QoR-40) before and 1 day after breast cancer surgery. MAIN OUTCOME MEASURES
  Other Names: PECs nerve injection
  Arms: PECs block group
Procedure: Sham block — Female undergone mastectomy and have received conventional analgesic methods
  Other Names: Non PECs block
  Arms: Non PECs block group

SUMMARY:
Impact of pectoral nerve block on postoperative pain and quality of recovery in patients undergoing breast cancer surgery: A prospective study

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy in women; surgery is still the mainstay for the treatment of breast cancer .

Postoperative pain can seriously reduce the quality of patient's life, and acute pain can even trigger chronic pain syndrome. Thoracic paravertebral, thoracic epidural, intercostal nerve, and interscalene brachial plexus blocks have been used for anesthesia and abirritation during mastectomy, but their applications are limited by the complicated technique of the procedures and several complications.

In recent years, there has been increasing interest on a novel, less invasive technique, the pectoral nerve (PECS) block. Numerous clinical trials have focused on the analgesic potential of the pectoral nerve block in breast augmentation surgery, small breast surgery, and breast cancer surgery, and have shown positive results.

Several prospective observational studies in recent years demonstrated that postoperative pain following breast surgery becomes chronic in up to 57% of women.

One of the most important risk factors is insufficiently treated postoperative acute pain. The current gold standard for acute postoperative pain is a preventive procedure-specific multimodal treatment including nonopioids, opioids and regional analgesia.

A recently published Cochran's meta-analysis demonstrated that regional analgesia [e.g. paravertebral block (PVB), local infiltration] might even reduce the risk of chronic postsurgical pain after breast surgery. According to a recently published guidelines, pectoral nerves (PECS) blocks seem to be an effective alternative to PVB to manage effectively postsurgical pain in major breast surgery.Anatomical studies revealed a different local anaesthetic spread following injections between the pectoralis major and minor muscles (PECS I) and a combination of the latter injection with a deeper injection between the pectoralis minor and serratus anterior muscles (PECS II) but the results were not conclusive. Many trials have been published and some meta-analyses revealed a high analgesic efficacy following PECS II blocks compared with no block or PVB.

However, one of these meta-analyses was criticised because of methodological problems (e.g. evidence assessment, missing sham block group), pain intensities not analysed separately for resting pain and pain during movement and comparisons with other established or emerging regional anaesthetic techniques (e.g. local infiltration, erector spinae block) were not performed.

ELIGIBILITY:
Inclusion Criteria:

1- all female planed for elective breast surgery

Exclusion Criteria:

1. Planned for bilateral axillary or bilateral reconstruction surgery.

   * Previous surgery on the surgical breast and/or axilla with the exception of partial mastectomy or sentinel lymph node biopsy Pre-existing pain in the axilla affecting the ability to use extremity for activities of daily living or requiring medication for treatment.
2. Current or past medical history of liver disease or cirrhosis with an elevated INR >1.4 or currently elevated transaminase levels.
3. known contraindications to peripheral nerve block placement.
4. Pregnant or breastfeeding.
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition
6. Planned additional surgery to the surgical breast or axilla in the next year (exception would be minor surgery to breast but not axilla such as simple tissue expander replacement or lumpectomy).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | 1year
  Postoperative pain score at rest Pain score using a verbal numerical scale (0-10) in one breast (bupivacaine) compared to the other breast (placebo).

SECONDARY OUTCOMES:
Patient's quality of life | 1 year
  1. Postoperative pain score on movement Pain score using a verbal numerical scale (0-10) in one breast (bupivacaine) compared to the other breast (placebo)
  2. Postoperative pain score at rest Pain score using a verbal numerical scale (0-10) in one breast (bupivacaine) compared to the other breast (placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Alaa eldin, Prof, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study will be available when the targeted number of cases reached
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: Full access
URL: http://ksa53516@gmail.com

REFERENCES:
- [Background] Ueshima H, Otake H, Hara E, Blanco R. How to Use Pectoral Nerve Blocks Effectively-An Evidence-Based Update. Asian J Anesthesiol. 2019 Jun 1;57(2):28-36. doi: 10.6859/aja.201906_57(2).0002. PMID 31382323
- [Background] Aarab Y, Ramin S, Odonnat T, Garnier O, Boissin A, Molinari N, Marin G, Perrigault PF, Cuvillon P, Chanques G. Pectoral Nerve Blocks for Breast Augmentation Surgery: A Randomized, Double-blind, Dual-centered Controlled Trial. Anesthesiology. 2021 Sep 1;135(3):442-453. doi: 10.1097/ALN.0000000000003855. PMID 34195767
- [Background] Daniel Pereira D, Bleeker H, Malic C, Barrowman N, Shadrina A. Pectoral nerve block and acute pain management after breast reduction surgery in adolescent patients. Can J Anaesth. 2021 Oct;68(10):1574-1575. doi: 10.1007/s12630-021-02037-8. Epub 2021 Jun 3. No abstract available. PMID 34081262